CLINICAL TRIAL: NCT05093192
Title: Characterising Tumour and Immune Cell Mobilisation Into Blood in Response to Acute Exercise in Chronic Lymphocytic Leukaemia
Brief Title: Mobilising Tumour and Immune Cells Via Exercise in Chronic Lymphocytic Leukaemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: Royal United Hospitals Bath NHS Foundation Trust (Other); University of Southampton (Other); Great Western Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, John Campbell, Principal Investigator, University of Bath
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 272493
Record Dates: First submitted 2021-09-06; First posted 2021-10-26 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Chronic Lymphocytic Leukemia; Minimal Residual Disease
Keywords: Exercise; Immunotherapy; Lymphocytes; ADCC
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasm, Residual; Motor Activity

STUDY DESIGN:
Intervention Model Description: A pilot, single-centre, Phase I trial containing 3 groups during different phases of CLL survivorship:
  * Cohort 1 (Pre treatment) CLL patients with asymptomatic early-stage disease monitored without anti-CLL treatment.
  * Cohort 2 (Treatment) Treatment eligible CLL patients receiving first-line anti-CLL treatment or patients receiving anti-CLL maintenance treatment.
  * Cohort 3 (Post treatment) CLL patients in complete remission (CR), complete remission with incomplete marrow recovery (CRi) or partial remission (PR) for at least 6 months following the completion of anti-CLL treatment.
  All participants will complete the study intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Pre-treatment CLL (Experimental): This group comprises patients who are diagnosed with CLL, but are asymptomatic and not receiving anti-CLL treatments (e.g. watch-and-wait disease).
  Interventions: Other: Exercise trial
- Cohort 2: During treatment CLL (Experimental): This group comprises patients who are diagnosed with CLL, have symptomatic disease, and are undergoing anti-CLL treatments (e.g. chemo-immunotherapy).
  Interventions: Other: Exercise trial
- Cohort 3: Post-treatment CLL (Experimental): This group comprises patients who were diagnosed with CLL, but are considered to be in either complete or partial remission following anti-CLL treatment for at least 6-months.
  Interventions: Other: Exercise trial

INTERVENTIONS:
Other: Exercise trial — Participants will perform a supervised acute bout of aerobic exercise over 20-30 minutes, corresponding to a target power output at an intensity +10 to 15% above ventilatory threshold.

SUMMARY:
Chronic lymphocytic leukaemia (CLL) is the most common adult blood cancer in the United Kingdom. CLL means that many cancer cells appear in the blood, bone marrow and other tissues, for example, the spleen where some blood cells reside. Most patients with CLL have been diagnosed by chance, have no symptoms as a result of CLL, and do not need urgent treatment. However, when the cancer cells build up, people experience symptoms of CLL, and treatment is required. One of the current treatments for CLL is chemo-immunotherapy, that targets and kills cancer cells in the blood. However, this treatment does not kill all cancer cells. Some cancer cells survive by 'hiding' in the bone marrow and tissues, like the spleen, where the treatment cannot get to, this is called minimal residual disease (MRD). MRD eventually builds up and patients experience symptoms of CLL again. New approaches to detect and treat MRD are needed. Research has shown, that the number of blood cells, increases after exercise and that many of these blood cells come from the bone marrow and other tissues.

This study will investigate if exercise can move CLL cancer cells that are 'hiding' in the bone marrow and other tissues into the blood, thus improving the detection of MRD. By moving cancer cells into blood, the investigators also think this will improve the way chemo-immunotherapy works. In this study, the investigators will investigate the number of cancer and natural killer (NK) cells in the blood after exercise, in three different groups of people with CLL: before treatment; during treatment; and after treatment has finished.

DETAILED DESCRIPTION:
Whilst repeated cycles of anti-cluster of differentiation (CD)20 immunotherapy are effective at killing large numbers of chronic lymphocytic leukaemia (CLL) cells, in the peripheral blood circulation, minimal residual disease (MRD) persists diffusely in the bone marrow and secondary lymphoid organs such as the lymph nodes and spleen. This is thought to be for a number of reasons. Firstly, malignant cells sequestered in lymphoid compartments receive protection from their stromal microenvironment. For example, T cells, dendritic cells and macrophages release pro-proliferative and apoptosis-inhibiting signalling pathways, that prolong CLL survival. Consequently, CLL cells in lymphoid tissues are much less susceptible to anti-CD20 immunotherapy, than CLL cells trafficking in the blood. This may be because the circulating CLL cells are not embedded into a protective stromal microenvironment. Secondly, to exert antibody-dependent cellular cytotoxicity (ADCC; i.e., the primary mechanism of action elicited by anti-CD20 immunotherapy against CLL cells) NK cells need to express CD16, a molecule expressed by CD56dim NK cells. However, these potent NK cells are unable to traffic from blood, where NK cells are more abundant, to secondary lymphoid tissues, because NK cells lack lymphoid homing markers. Thus, CLL cells are able to 'hide' from NK cells in lymphoid tissue, ensuring their ongoing survival. In light of the pro-survival features of the CLL microenvironment, new approaches to detect and treat MRD are sought.

It has been repeatedly shown, in one of the most reproduced findings in human physiology, that immune cell frequency in the peripheral blood increases profoundly, by approximately 50-100%, during a bout of aerobic exercise of moderate to vigorous intensity. This response reflects a redistribution of immune cells from marginal pools in the blood vessels, as well as from lymphoid organs, such as the spleen, bone marrow and lymph nodes into the blood, driven by increased haemodynamic forces and increased levels of catecholamines during exercise. In response to increased levels of exercise-induced catecholamines, beta-2 adrenergic receptors on the cell surface of lymphocytes, induce detachment from the vascular endothelium, thus promoting the mobilisation of lymphocytes into the peripheral blood circulation, during a bout of exercise, returning to pre exercise values in the 1 hour following exercise. The migration of immune cells into blood is comprised of all major immune cell types, including neutrophils, monocytes and lymphocytes. Due to the adrenergic mechanisms responsible there is a preferential mobilisation of the subtypes with the highest expression of beta-2 adrenergic receptors on the cell surface. NK cells are the most exercise responsive T lymphocyte population, followed by CD8+ T cells, B cells and CD4+ T cells. B cells express beta-2 adrenergic receptors and are therefore susceptible to mobilisation via exercise-induced catecholamines. In healthy persons, B cell frequency is increased in blood by approximately 50-100% during various different types of exercise including, cycling, running, rowing and resistance exercise. Furthermore, a rodent model of acute psychological stress - which induces similar adrenergic responses as exercise - demonstrated a similar B cell mobilisation pattern. An additional rodent model observed that acute stressors appear to redirect B cells from the bone marrow, suggesting that the B cells mobilised in response to exercise may have been mobilised from lymphoid tissue. Given these changes to immune cell kinetics, exercise may be an effective means of mobilising CLL cells from diffuse lymphoid tissues into the peripheral blood circulation, which may, in turn, facilitate the detection of MRD in CLL.

This exercise-induced mobilisation of CLL cells from lymphoid tissues may also increase the efficacy of anti-CD20 immunotherapy. Indeed, this process may facilitate the removal of CLL cells from protective, pro-survival microenvironments into the blood circulation. CLL cells survive in lymphoid tissue receiving external signals from the microenvironment promoting growth and survival. Furthermore, CD16+ NK cells, the primary effector cell in ADCC, do not express lymphoid homing markers on their cell surface, and cannot traffic to the lymphoid tissue to elicit potent ADCC responses. Therefore, in order to improve the depth and efficacy of treatment with anti-CD20 monoclonal antibodies (mAb), strategies need to be explored that remove CLL cells from their protective stromal microenvironment within lymphoid tissues, and mobilise into the blood circulation where CLL cells will encounter NK cells capable of eliciting ADCC. Exercise has the potential to redistribute B cells, and exercise has also been shown to increase the frequency of CD16+ NK cells, by over 500% into the blood circulation. Therefore, exercise may mobilise both CLL cells from their protective microenvironment and large numbers of effector NK cells capable of ADCC into the blood circulation, simultaneously. Thus, this process has the potential to improve the depth and efficacy of anti-CD20 mAb treatment.

It is of importance to examine the effects of exercise on CLL and CD16+ NK cells at different stages of the CLL survivorship. For instance, people with watch and wait CLL, who have not yet received anti-CLL therapy, enables investigations into the impact of exercise on both CLL tumour cell and immune cell kinetics, without the presence of confounding variables like anti-CLL treatments, or disease associated morbidities. Indeed, people with watch and wait CLL have no disease symptoms and are thus likely to have fewer contra-indications to exercise than CLL patients later in the CLL survivorship continuum.

Investigating the impact of exercise in people receiving anti-CLL treatments is also warranted, as those likely to benefit from the adjuvant effects of exercise on immunotherapy are, by reason, patients undergoing cycles of immunotherapy treatment. Thus, it is essential to explore how acute exercise is tolerated in people undergoing cycles of treatment, and assessment of the safety and acceptability of exercise is warranted. Moreover, chemoimmunotherapy induces immune-suppression which may nullify the immune changes induced by exercise. Accordingly, investigation of the effects of exercise on immune cell kinetics, as well as residual CLL tumour cells, is warranted in people receiving anti-CLL chemoimmunotherapy.

Lastly, examining the impact of exercise in people in CLL remission, following completion of anti-CLL treatment, is required as any exercise induced mobilisation of CLL cells may also facilitate the detection of MRD following anti-CLL treatment. Several studies have demonstrated that patients who achieved a clinical complete remission (CR) but with detectable MRD, can experience a disease relapse due to expansion of the residual CLL cells. Patients with CLL who achieve undetectable MRD (<1 CLL cell per 10,000 leukocytes in blood or bone marrow), following anti-CLL treatment have better clinical outcomes than those with detectable MRD. A meta-analysis of eleven international studies with a total of 2457 patients observed that undetectable MRD status after treatment with chemotherapy or chemoimmunotherapy in newly diagnosed CLL is associated with overall and progression free survival. Therefore, MRD is a robust post-treatment prognostic biomarker of tumour burden, required for predicting disease recurrence. However, due to the multicompartmental nature of CLL, the bone marrow and secondary lymphoid tissue may serve as reservoirs for residual disease. Therefore, exercise may be utilised to facilitate the detection of MRD by mobilising CLL cells from diffuse sites into the blood circulation, thus potentially accelerating the identification of disease progression in patients following anti-CLL treatment. It is also important to assess immune competency in people in remission following completion of anti-CLL therapy, as any immune suppression at this time may hinder any effects of exercise.

The hypotheses of this pilot study are as follows:

* An acute bout of exercise will increase the frequency of CLL tumour cells in the peripheral blood of people with CLL at different stages of CLL survivorship.
* An acute bout of exercise will increase the frequency of immune cells (e.g., CD16+ NK cells) in the peripheral blood of people with CLL at different stages of CLL survivorship.
* Exercise induced mobilisation of immune cells (e.g., NK cells) will improve the efficacy of anti-CD20 immunotherapy against CLL cells ex vivo.

ELIGIBILITY:
Cohort 1 (Pre Treatment)

Inclusion criteria:

* A diagnosis of: Chronic lymphocytic leukaemia. Defined by the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) guidelines as the presence of 5000 B cells per µL of peripheral blood, sustained for at least 3 months and confirmed by the blood smear, immunophenotype and in some cases genetic features of lymphoid cells.
* Age > 18 years old.
* Asymptomatic early-stage disease monitored without anti-CLL treatment.

Cohort 2 (Treatment)

Inclusion criteria:

* A diagnosis of: Chronic lymphocytic leukaemia. Defined by iwCLL guidelines as the presence of 5000 B cells per µL of peripheral blood, sustained for at least 3 months and confirmed by the blood smear, immunophenotype and in some cases genetic features of lymphoid cells.
* Age > 18 years old.
* Evidence of active disease defined as the following by the iwCLL guidelines:

  * Evidence of progressive marrow failure-the development of, or worsening of, anaemia and/or thrombocytopenia (in some patients, platelet counts <100 × 109/L may remain stable over a long period; this does not automatically require therapeutic intervention). Cut-off levels of haemoglobin less than 10 g/dL or platelet counts less than 100 × 109/L are generally regarded as an indication for treatment.
  * Massive (i.e., ≥6 cm below the left costal margin), progressive, or symptomatic splenomegaly.
  * Massive nodes (i.e., ≥10 cm in longest diameter), progressive, or symptomatic lymphadenopathy.
  * Progressive lymphocytosis with an increase of 50% or more over a 2-month period, or lymphocyte-doubling time (LDT) less than 6 months. LDT can be obtained by linear regression extrapolation of absolute lymphocyte counts obtained at intervals of 2 weeks over an observation period of 2 to 3 months; patients with initial blood lymphocyte counts less than 30 × 109/L may require a longer observation period to determine the LDT. Factors contributing to lymphocytosis other than CLL (e.g., infections or steroid administration) should be excluded.
  * Autoimmune complications, including anaemia or thrombocytopenia that respond poorly to corticosteroids.
  * Symptomatic or functional extranodal involvement (e.g., skin, kidney, lung, or spine). Disease-related symptoms defined as any of the following:

    * Unintentional weight loss of 10% or more within the previous 6 months.
    * Significant fatigue (i.e., Eastern Cooperative Oncology Group performance scale 2 or worse, cannot work, or unable to perform usual activities).
    * Fevers of 38.0°C or higher for 2 or more weeks without evidence of infection.
    * Night sweats for at least 1 month without evidence of infection.
* Recently initiated first-line treatment on one of the following regimes:

  * Fludarabine, cyclophosphamide and rituximab (FCR)
  * Ibrutinib monotherapy (I)
  * Ibrutinib + venetoclax (I+V)
  * Obinutuzumab + chlorambucil (O+C)
  * Bendamustine + rituximab (B+R)
  * Chlorambucil + ofatumumab (C+O)
  * Idelalisib + rituximab (I+R)
  * Venetoclax + rituximab (V+R)
  * Obinutuzumab monotherapy
  * Rituximab monotherapy
  * Ofatumumab monotherapy
  * Rituximab and chlorambucil
  * Chlorambucil monotherapy
* Ibrutinib or venetoclax maintenance treatment despite achieving complete remission (CR), complete remission with incomplete marrow recovery (CRi) or partial remission (PR).

Cohort 3 (Post treatment)

Inclusion criteria:

* A diagnosis of: Chronic lymphocytic leukaemia. Defined by iwCLL guidelines as the presence of 5000 B cells per µL of peripheral blood, sustained for at least 3 months and confirmed by the blood smear, immunophenotype and in some cases genetic features of lymphoid cells.
* Age > 18 years old.
* Complete remission (CR), complete remission with incomplete marrow recovery (CRi) or partial remission (PR) for at least 6 months following the completion of anti- CLL treatment.

Exclusion criteria:

* World Health Organisation (WHO)/ Eastern Cooperative Oncology Group (ECOG) performance status >1
* Pregnancy
* Deemed unsafe to exercise according to the Physical Activity Readiness Questionnaire (PARQ)
* Any comorbidity that is likely to progress or be exacerbated over the course of the trial period (e.g. history of syncopal events, significant cardiac or respiratory events)
* Cognitive impairment deemed a risk by the healthcare team for participation in the trial (e.g. diagnosis of neurodegenerative disease)
* Unable to understand explanations and/or provide informed consent
* Any condition and/or behaviour that would pose undue personal risk or introduce bias into the trial
* Following first-line treatment failure, patients with progressive disease or stable disease, as defined by iwCLL guidelines and described in Table 1 above.
* Recent b0lood counts at levels that are deemed to pose undue risk by the healthcare team.
* Any participant that has not received double coronavirus vaccinations, at least 14-days prior to the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Investigate whether an acute bout of exercise changes the frequency of CLL cells in peripheral blood. | Change from baseline CLL cell frequency to following 20-30 minutes of cycling.
  Number of CLL cells per microlitre will be measured by flow cytometry.

SECONDARY OUTCOMES:
Investigate whether an acute bout of exercise changes the frequency of immune cells (e.g., CD16+ NK cells), in peripheral blood. | Change from baseline immune cell frequency to following 20-30 minutes of cycling.
  Number of immune cells per microlitre will be measured by flow cytometry.
Investigate whether an acute bout of exercise changes the efficacy of anti-CD20 treatments against a CD20+ cell line or primary CLL cells. | Change from baseline CD20+ cell lysis to following 20-30 minutes of cycling.
  The percentage of CD20+ cell lysis will be measured using an ex vivo antibody-dependent cellular cytotoxicity assay.
Investigate whether an acute bout of exercise changes whole blood counts. | Change from baseline whole blood counts to following 20-30 minutes of cycling.
  Whole blood counts, in cells per litre.
Investigate whether an acute bout of exercise changes immunoglobulins. | Change from baseline immunoglobulins to following 20-30 minutes of cycling.
  Immunoglobulins, in ng/mL, measured by enzyme-linked immunosorbent assay (ELISA).
Investigate whether an acute bout of exercise changes serum C1q. | Change from baseline C1q to following 20-30 minutes of cycling.
  C1q, in ng/mL, measured by ELISA.
Investigate whether an acute bout of exercise changes serum C3. | Change from baseline C3 to following 20-30 minutes of cycling.
  C3, in ng/mL, measured by turbidimetry.
Investigate whether an acute bout of exercise changes plasma C-reactive protein (CRP). | Change from baseline CRP to following 20-30 minutes of cycling.
  CRP, in pg/mL, measured by turbidimetry.
Investigate whether an acute bout of exercise changes capillary glucose. | Change from baseline glucose to following 20-30 minutes of cycling.
  Glucose, in mmol/L, measured by an Abbot blood glucose meter.
Investigate whether an acute bout of exercise changes capillary lactate. | Change from baseline lactate to following 20-30 minutes of cycling.
  Lactate, in mmol/L, measured by a blood lactate meter.

OTHER OUTCOMES:
Differences in physical fitness amongst groups along CLL survivorship spectrum. | Baseline, pre-intervention.
  Ventilatory threshold, in mL/kg/min, will be measured by a submaximal exercise test.
Differences in height amongst groups along CLL survivorship spectrum. | Baseline, pre-intervention.
  Height, in centimetres, will be measured by a stadiometer.
Differences in weight amongst groups along CLL survivorship spectrum. | Baseline, pre-intervention.
  Weight, in kilograms, will be measured by an electronic weighing scale.
Differences in fat mass amongst groups along CLL survivorship spectrum. | Baseline, pre-intervention.
  Fat mass, in kilograms, will be measured by Bioelectrical Impedance Analysis (BIA).
Differences in lean mass amongst groups along CLL survivorship spectrum. | Baseline, pre-intervention.
  Lean mass, in kilograms, will be measured by BIA.
Differences in waist-to-hip circumference amongst groups along CLL survivorship spectrum. | Baseline, pre-intervention.
  Waist-and-hip circumference, as a ratio.
Differences in physical activity amongst groups along CLL survivorship spectrum. | Baseline, pre-intervention.
  Physical activity, in hours per day, will be measured by the International Physical Activity Questionnaire.
Differences in stress amongst groups along CLL survivorship spectrum. | Baseline, pre-intervention.
  Stress, in a scale of 0-4, will be measured by the Perceived Stress Scale.
Differences in fatigue amongst groups along CLL survivorship spectrum. | Baseline, pre-intervention.
  Fatigue, in a 5-point scale of 'not at all' to 'very much', will be measured by the Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale.
Differences in sleep amongst groups along CLL survivorship spectrum. | Baseline, pre-intervention.
  Sleep, in a scale of 0-3, will be measured by the Pittsburgh Sleep Quality Index.
Differences in quality of life amongst groups along CLL survivorship spectrum. | Baseline, pre-intervention.
  Quality of life, in a scale of 1-4, will be measured by the Health-Related Quality of Life questionnaire.
Differences in blood pressure amongst groups along CLL survivorship spectrum. | Baseline, pre-intervention.
  Blood pressure, in mmHg, will be measured by an automated blood pressure cuff.
Differences in viral infection history amongst groups along CLL survivorship spectrum. | Baseline, pre-intervention.
  Viral infection history, in a 4-point scale of 'not at all' to 'very much', will be measured by questionnaire.
Quantification of CLL cells in adipose tissue in groups with watch-and-wait or recessive CLL. | Baseline, pre-intervention.
  Number of CLL cells per microgram of adipose tissue will be measured by flow cytometry.
Determination of the safety of exercise amongst groups along CLL survivorship spectrum. | Through the cycling intervention, averaging 20-30 minutes of cycling.
  Quantified by the incidence of adverse events.
Determination of the feasibility of exercise amongst groups along CLL survivorship spectrum. | Through the cycling intervention, averaging 20-30 minutes of cycling.
  Quantified by the percentage difference between the prescribed and achieved exercise per session.
Determination of the uptake of exercise trials amongst groups along CLL survivorship spectrum. | Baseline, pre-intervention.
  Quantified by the percentage of participants who attend screening.
Determination of the retention of exercise trials amongst groups along CLL survivorship spectrum. | Through study completion, an average of 17-weeks.
  Quantified by the percentage of participants who complete all trial visits.

CONTACTS AND LOCATIONS:
Overall Officials: John P Campbell, PhD, Principal Investigator — University of Bath
Locations (2):
- United Kingdom (2):
  - Royal United Hospital Bath NHS Foundation Trust, Bath, Bath & Northeast Somerset
  - University of Bath, Bath, Bath & Northeast Somerset

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/92/NCT05093192/ICF_000.pdf